CLINICAL TRIAL: NCT05642754
Title: Communicating Uncertainty About the Effects of Wearing Glasses to Reduce the Chance of Getting COVID (Corona Virus Disease): Protocol for a Randomized Trial
Brief Title: Glassy Trial for Effects of Wearing Glasses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trustees of Dartmouth College (Other)
Collaborators: Norwegian Institute of Public Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: 557972; CPHS 32615 (Other: Dartmouth College CPHS)
Record Dates: First submitted 2022-11-30; First posted 2022-12-08 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: COVID-19
Keywords: Colloquial language; uncertainty; bias
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: 3 options for describing bias/uncertainty about results 2 options for margin of error around main result (we will run the trial twice on 2 different online platforms)
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- GRADE + margin of error (Active Comparator): Overall uncertainty using GRADE* language AND margin of error around main result
  * Based on the Cochrane Effective Practice and Organisation of Care Group's guidance for communicating the certainty of evidence based on the Grading of Recommendations Assessment, Development and Evaluation (GRADE) approach to assessing the certainty of evidence
  Interventions: Other: Overall uncertainty language
- Colloquial language AND margin of error (Active Comparator): Colloquial language developed to describe overall study uncertainty AND margin of error around main result
  Interventions: Other: Overall uncertainty language
- No overall uncertainty language AND margin of error (Active Comparator): No overall uncertainty language AND margin of error around main result
  Interventions: Other: Overall uncertainty language
- GRADE -No margin of error (Active Comparator): Overall uncertainty using GRADE* language and NO margin of error around main result
  * Based on the Cochrane Effective Practice and Organisation of Care Group's guidance for communicating the certainty of evidence based on the Grading of Recommendations Assessment, Development and Evaluation (GRADE) approach to assessing the certainty of evidence
  Interventions: Other: Overall uncertainty language
- Colloquial - No margin of error (Active Comparator): Colloquial language developed to describe overall study uncertainty and NO margin of error around main result
  Interventions: Other: Overall uncertainty language
- No overall uncertainty language AND no margin of error (Placebo Comparator): No overall uncertainty language and NO margin of error around main result
  Interventions: Other: Overall uncertainty language

INTERVENTIONS:
Other: Overall uncertainty language — Researchers are testing different forms of information about overall study uncertainty and margin of error around main result
  Other Names: Margin of error around main result

SUMMARY:
Randomized trial testing 6 forms of a communication summarizing the results of a recent study (about the effects of wearing glasses on reducing covid infection risk).

The goal of the trial is to test the effect of different language options to describe uncertainty, and of including the margin of error around the main result.

DETAILED DESCRIPTION:
The study is designed as a proof-of-concept exercise to develop and test a communication meant to summarize the results of a recent randomized trial examining the effects of wearing glasses on the chance of developing COVID-19.

The objectives of the randomized trial are:

* To compare the effects of three ways of communicating the overall uncertainty of the effects of wearing glasses to reduce the chance of getting COVID and
* To compare the effects of including the margin of error (confidence interval) compared to not including it.

Researchers will conduct an online, parallel group, individually randomized, pragmatic trial using a 3x2 factorial design, ie, 3 uncertainly language options (GRADE language, colloquial language or none 2 options for the statistical margin of error for the main results (margin of error language or none).

ELIGIBILITY:
Inclusion Criteria:

* >= 18 years old
* literate in English or Norwegian
* currently residing in Norway or the United States

Exclusion Criteria:

* individuals who regularly wear any kind of glasses (i.e., prescription or sunglasses) all or most of the time

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 960 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
understanding of overall uncertainty of benefit (of wearing glasses to reduce the chance of covid infection) | within 1 day
  How sure about the effect (4 point scale from very unsure to very sure)
understanding of overall uncertainty of harm (of wearing glasses to reduce the chance of covid infection) | within 1 day
  How sure about the effect (4 point scale from very unsure to very sure)
sufficiency of what is known about the effects of wearing glasses to reduce the chance of covid infection | within 1 day
  How sure about the effect (4 point Likert scale)
Understanding the margin of error around the benefit of wearing glasses to reduce covid | within 1 day
  this is a co-primary outcome which will be used only to compare the 3 versions that include the margin of error to the 3 versions that do not

SECONDARY OUTCOMES:
perceived effect of wearing glasses to reduce chance of covid infection | within 1 day
  What is the effect on a 5 point scale (lowers a lot, lowers a little, no effect, increase a little, increases a lot
how likely is it that wearing glasses reduces the chance of covid infection | within 1 day
  4 point scale (very likely, likely, unlikely, very unlikely)
intended behavior (if there were a surge in covid in your area, how likely would you be to wear glasses to reduce the chance of covid infection | within 1 day
  4 point scale (very likely, likely, unlikely, very unlikely
intended behavior (if there were very few cases of covid in your area, how likely would you be to wear glasses to reduce the chance of covid infection | within 1 day
  4 point scale (very likely, likely, unlikely, very unlikely
perceptions fo information provided (trustworthy summary?) | within 1 day
  4 point Likert scale (strongly agree, agree, disagree, strongly disagree)
perceptions fo information provided (sufficient summary?) | within 1 day
  4 point Likert scale (strongly agree, agree, disagree, strongly disagree)
perceptions fo information provided (clarity of info about benefit) | within 1 day
  4 point scale (very clear, clear, unclear, very unclear)
perceptions fo information provided (clarity of info about harm) | within 1 day
  4 point scale (very clear, clear, unclear, very unclear)
perceptions fo information provided (info helpful?) | within 1 day
  4 point scale (very helpful, helpful, unhelpful, very unhelpful)
perceptions fo information provided (share info with others?) | within 1 day
  4 point scale (definitely yes, probably yes, probably no, definitely no)
Decisional conflict (hard to make decision) | within 1 day
  4 point LIkert scale (strongly agree, agree, disagree, strongly disagree)
Decisional conflict (made informed decision) | within 1 day
  4 point LIkert scale (strongly agree, agree, disagree, strongly disagree)
Decisional conflict (satisfied with decision) | within 1 day
  4 point LIkert scale (strongly agree, agree, disagree, strongly disagree)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Woloshin, MD, Principal Investigator — Dartmouth Institute for Health Policy and Clincal Practice; Andy Oxman, MD, Principal Investigator — Norwegian Institute of Public Health
Locations (1):
- Norwegian Institute of Public Health, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Holst C, Woloshin S, Oxman AD, Rose C, Rosenbaum S, Munthe-Kaas HM. Alternative Presentations of Overall and Statistical Uncertainty for Adults' Understanding of the Results of a Randomized Trial of a Public Health Intervention: Parallel Web-Based Randomized Trials. JMIR Public Health Surveill. 2025 Mar 18;11:e62828. doi: 10.2196/62828. PMID 40101228